CLINICAL TRIAL: NCT00076102
Title: Phase II Trial of Pirfenidone in Children, Adolescents, and Young Adults With Neurofibromatosis Type 1 and Progressive Plexiform Neurofibromas
Brief Title: Pirfenidone in Children and Young Adults With Neurofibromatosis Type I and Progressive Plexiform Neurofibromas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brigitte Widemann, M.D., Dr. Brigitte Widemann, M.D., National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040080; 04-C-0080; FD-R-0002128 (Other Grant/Funding Number: FDA OOPD); NCT00078936 (obsolete NCT alias)
Record Dates: First submitted 2004-01-13; First posted 2004-01-14 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Neurofibromatosis 1; Neurofibroma, Plexiform
Keywords: Side Effect; Oral Administration; Nerve Sheath Tumor; Antifibrotic Agent; Volumetric Tumor Measurement; Plexiform Neurofibroma; Neurofibromatosis Type 1; Volumetric MRI Analysis; Time to Progression; NF1
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Nerve Sheath Neoplasms | interventions — pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirfenidone (Experimental): Pirfenidone orally as capsules three times a day approximately every 8 hours for cycles of 28 days with no rest period between cycles (28 day treatment cycles); 500 mg/m^2 every 8 hours (1500 mg/m2/day).
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone orally as capsules three times a day approximately every 8 hours for cycles of 28 days with no rest period between cycles (28 day treatment cycles); 500 mg/m^2 every 8 hours (1500 mg/m2/day).
  Other Names: Esbriet; Deskar

SUMMARY:
Background:

Neurofibromatosis Type 1 (NF1) is an autosomal dominant, progressive genetic disorder characterized by diverse clinical manifestations. Patients with NF1 have an increased risk of developing tumors of the central and peripheral nervous system including plexiform neurofibromas, which are benign nerve sheath tumors that may cause severe morbidity and possible mortality. The histopathology of these tumors suggests that events connected with formation of fibroblasts might constitute a point of molecular vulnerability. Gene profile analysis demonstrates overexpression of fibroblast growth factor, epidermal growth factor, and platelet-derived growth factor in plexiform neurofibromas in patients with NF1. Pirfenidone is a novel antifibrotic agent that inhibits these and other growth factors. Clinical experience in adults has demonstrated that pirfenidone is effective in a variety of fibrosing conditions and pirfenidone is presently under study in a phase II trial for adults with progressive plexiform neurofibromas. A phase I trial of pirfenidone in children and young adults with NF1 and plexiform neurofibromas was completed, and has established the phase II dose (the dose resulting in a mean drug exposure [AUC] not more than 1 standard deviation below the mean drug exposure [AUC] in adults who received pirfenidone at the dose level demonstrating activity in fibrosing conditions). Pirfenidone has been well tolerated.

Objectives:

To determine whether pirfenidone increases the time to disease progression based on volumetric measurements in children and young adults with NF1 and growing plexiform neurofibromas.

To define the objective response rate to pirfenidone in NF1-related plexiform neurofibromas.

To describe and define the toxicities of pirfenidone.

Eligibility:

Individuals (greater than or equal to 3 years to less than or equal to 21 years of age) with a clinical diagnosis of NF1 and inoperable, measurable, and progressive plexiform neurofibromas that have the potential to cause substantial morbidity.

Design:

The phase II dose will be used in a single stage, single arm phase II trial The natural history of the growth of plexiform neurofibromas is unknown. For this reason, time to disease progression on the placebo arm of an ongoing National Cancer Institute (NCI) Pediatric Oncology Branch (POB) placebo-controlled, double-blind, cross-over phase II trial of the farnesyltransferase inhibitor R115777 for children and young adults with NF1 and progressive plexiform neurofibromas.

Funding source - Food and Drug Administration (FDA) Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
Background:

Neurofibromatosis Type 1 (NF1) is an autosomal dominant, progressive genetic disorder characterized by diverse clinical manifestations. Patients with NF1 have an increased risk of developing tumors of the central and peripheral nervous system including plexiform neurofibromas, which are benign nerve sheath tumors that may cause severe morbidity and possible mortality. The histopathology of these tumors suggests that events connected with formation of fibroblasts might constitute a point of molecular vulnerability. Gene profile analysis demonstrates overexpression of fibroblast growth factor, epidermal growth factor, and platelet-derived growth factor in plexiform neurofibromas in patients with NF1. Pirfenidone is a novel antifibrotic agent that inhibits these and other growth factors. Clinical experience in adults has demonstrated that pirfenidone is effective in a variety of fibrosing conditions and pirfenidone is presently under study in a phase II trial for adults with progressive plexiform neurofibromas. A phase I trial of pirfenidone in children and young adults with NF1 and plexiform neurofibromas was completed, and has established the phase II dose (the dose resulting in a mean drug exposure [AUC] not more than 1 standard deviation below the mean drug exposure [AUC] in adults who received pirfenidone at the dose level demonstrating activity in fibrosing conditions). Pirfenidone has been well tolerated.

Objectives:

To determine whether pirfenidone increases the time to disease progression based on volumetric measurements in children and young adults with NF1 and growing plexiform neurofibromas.

To define the objective response rate to pirfenidone in NF1-related plexiform neurofibromas.

To describe and define the toxicities of pirfenidone.

Eligibility:

Individuals (greater than or equal to 3 years to less than or equal to 21 years of age) with a clinical diagnosis of NF1 and inoperable, measurable, and progressive plexiform neurofibromas that have the potential to cause substantial morbidity.

Design:

The phase II dose will be used in a single stage, single arm phase II trial The natural history of the growth of plexiform neurofibromas is unknown. For this reason, time to disease progression on the placebo arm of an ongoing National Cancer Institute (NCI) Pediatric Oncology Branch (POB) placebo-controlled, double-blind, cross-over phase II trial of the farnesyltransferase inhibitor R115777 for children and young adults with NF1 and progressive plexiform neurofibromas will be used as historical control to determine if pirfenidone increases time to disease progression. Eligibility criteria and method of tumor measurements are identical for both trials.

Pirfenidone will be administered orally as capsules at a dose of 500 mg/m^2 three times a day (q8h) for cycles of 28 days with no rest period between cycles based on the results of our pediatric phase I trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: greater than or equal to 3 years and Less than or equal to 21 years of age. Required body surface area (BSA): greater than or equal to 0.31 m^2.
  2. Diagnosis: Patients with NF1 and progressive plexiform neurofibromas that have the potential to cause significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or significant cosmetic problems, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings, but should be considered if malignant degeneration of a plexiform neurofibroma is clinically suspected. In addition to plexiform neurofibroma(s), all study subjects must have at least one other diagnostic criteria for NF1 listed below (National Institutes of Health (NIH) Consensus Conference):

  <!-- -->

  1. Six or more cafe-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects)
  2. Freckling in the axilla or groin
  3. Optic glioma
  4. Two or more Lisch nodules
  5. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  6. A first-degree relative with NF1

In this study a plexiform neurofibroma is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal plexiform neurofibroma involves two or more levels with connection between the levels or extending laterally along the nerve.

3. Measurable disease: Patients must have measurable plexiform neurofibroma(s). For the purpose of this study a measurable lesion will be defined as a lesion of at least 3 cm measured in one dimension. There must be evidence of recurrent or progressive disease as documented by an increase in size or the presence of new plexiform neurofibromas on MRI. Progression at the time of study entry is defined as:

A. A measurable increase of the plexiform neurofibroma (greater than or equal to 20% increase in the volume, or a greater than or equal to 13% increase in the product of the two longest perpendicular diameters, or a greater than or equal to 6% increase in the longest diameter) over the last two consecutive scans (magnetic resonance imaging (MRI) or computed tomography (CT), or over the time period of approximately one year prior to evaluation for this study.

B. Patients who underwent surgery for a progressive plexiform neurofibroma will be eligible to enter the study after the surgery, provided the plexiform neurofibroma was incompletely resected and is measurable.

4. Prior therapy: Patients with NFI are eligible at the time of recurrence or progression of an inoperable plexiform neurofibroma. Patients will only be eligible if complete tumor resection is not feasible, or if a patient with a surgical option refuses surgery.

Since there is no standard effective chemotherapy for patients with NF1 and progressive plexiform neurofibromas, patients may be treated on this trial without having received prior medical therapy.

Patients who received prior medical treatment for their plexiform neurofibroma(s) must have recovered from the toxic effects of all prior therapy before entering this study. The Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE-3) Version 3.0 will be used for toxicity assessment. A copy of the CTCAE version 3.0 can be downloaded from the CTEP home page (http:// ctep.cancer.gov). Recovery is defined as a toxicity grade less than 2, unless otherwise specified in the Inclusion and Exclusion Criteria.

Patients must have had their last dose of radiation therapy at least six weeks prior to study entry, and their last dose of chemotherapy at least four weeks prior to study entry. Patients who received G-CSF after the prior cycle of chemotherapy must be off G-CSF for at least one week prior to entering this study.

5. Performance Status: Performance Status: Patients should have a life expectancy of at least 12 months. Patients greater than 10 years must have a Karnofsky performance level greater than or equal to 50, and children less than or equal to 10 years must have a Lansky performance level greater than or equal to 50. Patients who are wheelchair bound because of paralysis should be considered ambulatory when they are up in their wheel chair.

6. Hematologic Function: Patients must have an absolute granulocyte count greater than or equal to 1,500/uL, a hemoglobin greater than or equal to 9.0 gm/dl, and a platelet count greater than or equal to 150,000/microliter at study entry (all transfusion independent).

7. Hepatic Function: Patients must have a bilirubin within normal limits and serum glutamic pyruvic transaminase (SGPT) less then or equal to 2x upper limit of normal. Patients with Gilbert syndrome are excluded from the requirement of a normal bilirubin. (Gilbert syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis).

8. Renal Function: Patients must have an age-adjusted normal serum creatinine (see table below) OR a creatinine clearance greater than or equal to 70 mL/min/1.73 m^2.

Age Maximum Serum Creatinine

(years) (mg/dl)

less than or equal to 5 0.8

5 less than age less than or equal to 10 1.0

10 less than age less than or equal to 15 1.2

greater than 15 1.5

9. Informed Consent: All patients or their legal guardians (if the patients is less than 18 years old) must sign an Institutional Review Board (IRB) approved document of informed consent (screening protocol) prior to performing studies to determine patient eligibility. After confirmation of patient eligibility all patients or their legal guardians must sign the protocol specific informed consent to document their understanding of the investigational nature and the risks of this study before any protocol related studies are performed (other than the studies which were performed to determine patient eligibility). When appropriate, pediatric patients will be included in all discussions. Age appropriate assent forms for children from 7 through 12 years, and for children from 13 through 17 years have been developed and will be signed by the pediatric patients, when appropriate, in order to obtain written assent.

10. Durable Power of Attorney (DPA): All patients greater than or equal to 18 years of age will be offered the opportunity to assign DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

11. Patients must be able to take pirfenidone by mouth. Capsules can be opened and content mixed with food for easier consumption in small children.

12. Patients (both male and female) must be willing to practice birth control (including abstinence) during and for two months after treatment, if of a child-bearing age. For purposes of the protocol, all patients greater than 9 years of age or those showing pubertal development will be considered of childbearing age.

13. Ability to undergo magnetic resonance imaging (MRI) and no contraindication for MRI examinations following the MRI protocol outlined.

EXCLUSION CRITERIA:

1. Pregnant or breast feeding females are excluded, because the toxic effects and pharmacology of pirfenidone in the fetus and newborn are unknown.
2. Clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate pirfenidone or are likely to interfere with the study procedures or results.
3. An investigational agent within the past 30 days.
4. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, immunotherapy, or biologic therapy (for example interferon).
5. Inability to return for follow-up visits or obtain follow-up studies required to assess toxicity and response to therapy.
6. Prior treatment with pirfenidone.
7. Evidence of an optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07-21 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Memorial Hospital, Chicago, Chicago, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Childrens Hospital, Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital, Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cain WC, Stuart RW, Lefkowitz DL, Starnes JD, Margolin S, Lefkowitz SS. Inhibition of tumor necrosis factor and subsequent endotoxin shock by pirfenidone. Int J Immunopharmacol. 1998 Dec;20(12):685-95. doi: 10.1016/s0192-0561(98)00042-3. PMID 9877280
- [Background] DeClue JE, Heffelfinger S, Benvenuto G, Ling B, Li S, Rui W, Vass WC, Viskochil D, Ratner N. Epidermal growth factor receptor expression in neurofibromatosis type 1-related tumors and NF1 animal models. J Clin Invest. 2000 May;105(9):1233-41. doi: 10.1172/JCI7610. PMID 10791998
- [Background] Evans DG, Baser ME, McGaughran J, Sharif S, Howard E, Moran A. Malignant peripheral nerve sheath tumours in neurofibromatosis 1. J Med Genet. 2002 May;39(5):311-4. doi: 10.1136/jmg.39.5.311. PMID 12011145
- [Result] Widemann BC, Babovic-Vuksanovic D, Dombi E, Wolters PL, Goldman S, Martin S, Goodwin A, Goodspeed W, Kieran MW, Cohen B, Blaney SM, King A, Solomon J, Patronas N, Balis FM, Fox E, Steinberg SM, Packer RJ. Phase II trial of pirfenidone in children and young adults with neurofibromatosis type 1 and progressive plexiform neurofibromas. Pediatr Blood Cancer. 2014 Sep;61(9):1598-602. doi: 10.1002/pbc.25041. Epub 2014 Apr 22. PMID 24753394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 participants were enrolled in this study
Period: Overall Study
Arm/Group | Pirfenidone
Started | 36
Completed | 31
Not Completed | 5
Not completed — Clinical progression | 1
Not completed — Progression in pre-existing brain tumor | 1
Not completed — plexiform neurofibroma surgery | 1
Not completed — refusal of further therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pirfenidone
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.81 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Disease Progression
Description: Time to progression is defined as greater than or equal to 20% increase in plexiform neurofibromas (PN) volume on magnetic resonance imaging (MRI).
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pirfenidone
Number analyzed (Participants) | 36
Months | 13.2 [8.2 to 18.6]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Pirfenidine: Pirfenidone orally as capsules three times a day approximately every 8 hours for cycles of 28 days with no rest period between cycles (28 day treatment cycles); 500 mg/m^2 every 8 hours (1500 mg/m2/day).
Arm/Group | Pirfenidine
Number analyzed (Participants) | 36
Participants | 36

3. Primary Outcome: Percentage of Participants Who Had an Objective Response Rate
Description: Objective response rate is defined as a complete response (CR) or partial response (PR). Complete response is a complete resolution of all measurable or palpable soft tissue tumors for ≥4 weeks and no appearance of new lesions. Partial response is a ≥50% reduction in the sum of the volume of all index lesions for ≥4 weeks.
Time Frame: ≥4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Pirfenidine
Number analyzed (Participants) | 31
percentage of participants
  Complete Response | 0
  Partial Response | 0

4. Secondary Outcome: Quality of Life (QOL) Using the Impact of Pediatric Illness (IPI) Scale at Baseline
Description: Quality of life was assessed by the Impact of Pediatric Illness scale for children 6-18 years of age. The child's primary caregiver completed the proxy Parent Form and children answered either the self-report Child or Adolescent (11-18 years) Form. The parallel IPI Scale forms assess four domains: adaptive behavior, emotional functioning, medical/physical status, and cognitive functioning. Responses to the 43 items are made on a 3-or5-point Likert scale (1 to 5 for Parent and Adolescent Form and 1, 3, 5 for the Child Form) ranging from "not at all" to "a lot". Item scores are transformed to a scale of 0-100, and then mean scores are calculated for the four domains and total scale with higher scores indicating better QOL. Baseline comparisons between child and parent total and domain scores were performed.
Time Frame: Baseline
Population: Of the 36 patients enrolled, 28 were within the age range of the IPI Scale at baseline. Two patients did not have any QOL forms completed; one did not have a baseline evaluation, and six patients had missing follow-up evaluations. Thus, QOL data is presented for 19 subjects.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pirfenidine
Number analyzed (Participants) | 19
Scores on a scale
  Total score parent | 72.7 (10.7)
  Total score child | 69.1 (12.0)
  Parent proxy-adaptive behavior | 72.1 (10.2)
  Child Self-Report-adaptive behavior | 76.7 (11.8)
  Parent proxy - emotional functioning | 72.4 (13.4)
  Child Self-Report-emotional functioning | 63.7 (14.7)
  Parent proxy - medical/physical status | 77.6 (15.1)
  Child Self-Report - medical/physical status | 67.1 (16.2)
  Parent proxy - cognitive functioning | 62.9 (19.6)
  Child Self-Report- cognitive functioning | 69.4 (18.5)
Statistical Analysis 1: Comparison: Pirfenidine; F=5.45 under the null hypothesis; Test type: Other; p = 0.0301, ANOVA — The reported F statistic and p-value are representative of the difference in the Parent proxy Form and the Child Self-Report Form response for Adaptive Behavior
Statistical Analysis 2: Comparison: Pirfenidine; F = 6.56 under the null hypothesis; Test type: Other; p = 0.0186, ANOVA — The reported p-value is representative of the difference in the Parent proxy Form and the Child Self-Report Form response for Emotional Functioning
Statistical Analysis 3: Comparison: Pirfenidine; F=11.23 under the null hypothesis; Test type: Other; p = 0.0032, ANOVA — The reported p-value is representative of the difference in the Parent proxy Form and the Child Self-Report Form response for Medical/Physical Status

5. Secondary Outcome: Longitudinal Total Quality of Life Scores Assessed by the Impact of Pediatric Illness Scale
Description: Quality of life was assessed by the Impact of Pediatric Illness scale for children 6-18 years of age. The child's primary caregiver completed the proxy Parent Form and children answered either the self-report Child or Adolescent (11-18 years) Form prior to cycles 1, 4, 7 and 10. The parallel IPI Scale forms assess four domains: adaptive behavior, emotional functioning, medical/physical status, and cognitive functioning. Responses to the 43 items are made on a 3-or5-point Likert scale (1 to 5 for Parent and Adolescent Form and 1, 3, 5 for the Child Form) ranging from "not at all" to "a lot". Item scores are transformed to a scale of 0-100, and then mean scores are calculated for the four domains and total scale with higher scores indicating better QOL.
Time Frame: prior to cycles 1, 4, 7 and 10.
Population: Of the 36 pts enrolled, 28 were within the age range of the IPI Scale at baseline. 2 pts did not have any QOL forms completed; 1 did not have a baseline & 6 pts had missing f/u evals. QOL data is presented for 19 pts. Due to pts not completing forms at random f/u evals, some time points have fewer than 19 pts included in the longitudinal analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pirfenidine
Number analyzed (Participants) | 19
scores on a scale
  Parent Baseline (to Cycle 4) | 71.1 (13.1)
  Parent Pre Cycle 4 | 71.8 (10.7)
  Child Baseline (to Cycle 4) | 67.9 (12.9)
  Child Pre Cycle 4 | 69.8 (10.8)
  Parent Baseline (to Cycle 7): number analyzed (Participants) | 16
  Parent Baseline (to Cycle 7) | 71.7 (11.5)
  Parent Pre Cycle 7: number analyzed (Participants) | 17
  Parent Pre Cycle 7 | 70.6 (9.0)
  Child Baseline (to Cycle 7): number analyzed (Participants) | 16
  Child Baseline (to Cycle 7) | 69.5 (12.8)
  Child Pre Cycle 7: number analyzed (Participants) | 17
  Child Pre Cycle 7 | 71.4 (12.3)
  Parent Baseline (to Pre Cycle 10): number analyzed (Participants) | 13
  Parent Baseline (to Pre Cycle 10) | 71.56 (12.6)
  Parent Pre Cycle 10: number analyzed (Participants) | 15
  Parent Pre Cycle 10 | 72.1 (7.8)
  Child Baseline (to Pre Cycle 10): number analyzed (Participants) | 13
  Child Baseline (to Pre Cycle 10) | 67.5 (13.0)
  Child Pre Cycle 10: number analyzed (Participants) | 15
  Child Pre Cycle 10 | 68.3 (14.1)
Statistical Analysis 1: Comparison: Pirfenidine; F=0.25 under the null hypothesis; Test type: Other; p = 0.6263, ANOVA
Statistical Analysis 2: Comparison: Pirfenidine; F= 0.87 under the null hypothesis; Test type: Other; p = 0.3625, ANOVA
Statistical Analysis 3: Comparison: Pirfenidine; F=0.31 under the null hypothesis; Test type: Other; p = 0.5877, ANOVA
Statistical Analysis 4: Comparison: Pirfenidine; F=1.27 under the null hypothesis; Test type: Other; p = 0.2767, ANOVA
Statistical Analysis 5: Comparison: Pirfenidine; F=0.04 under the null hypothesis; Test type: Other; p = 0.8466, ANOVA
Statistical Analysis 6: Comparison: Pirfenidine; F=0.18 under the null hypothesis; Test type: Other; p = 0.6774, ANOVA

6. Secondary Outcome: Number of Participants With A Response Evaluation Determined by the Comparison of One-Dimensional (1D) Magnetic Resonance Imaging
Description: Index lesions will be followed for progression by 1D magnetic resonance imaging. Progression is defined as a ≥20% increase in the volume of at least one of the index plexiform neurofibromas compared to the pretreatment volume measured prior to the start of treatment.
Time Frame: Prior to cycles 1, 4, 7, and 10 and then every 6 cycles thereafter until progression
Population: This outcome measure was not done because only 3D imaging was performed. Due to a detailed comparison of 1D-2D and 3D imaging for another study (Tipifarnib R115777) the investigator determined that a detailed comparison of 1D-2D and 3D analysis would really add no new knowledge. Therefore only 3D analysis was performed for this trial.
Arm/Group | Pirfenidone
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With A Response Evaluation Determined by the Comparison of Two-Dimensional (2D) Magnetic Resonance Imaging
Description: Index lesions will be followed for progression by 2D magnetic resonance imaging. Progression is defined as a ≥20% increase in the volume of at least one of the index plexiform neurofibromas compared to the pretreatment volume measured prior to the start of treatment.
Time Frame: Prior to cycles 1, 4, 7, and 10 and then every 6 cycles thereafter until progression
Population: as for outcome 6
Arm/Group | Pirfenidone
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With A Response Evaluation Determined by the Comparison of Three-Dimensional (3D) Magnetic Resonance Imaging
Description: Index lesions will be followed for progression by 3D magnetic resonance imaging. Compete response is a complete resolution of all measurable or palpable soft tissue tumors for ≥4 weeks and no appearance of new lesions. Partial response is a ≥50% reduction in the sum of the volume of all index lesions for ≥4 weeks. Progression is defined as a ≥20% increase in the volume of at least one of the index plexiform neurofibromas compared to the pretreatment volume measured prior to the start of treatment. Stable disease is a <20% increase, and <25% decrease in the sum of the volume of all index lesions for ≥4 weeks. Minor response is a ≥25% but <50% reduction in the sum of the volume of all index lesions for ≥4 weeks.
Time Frame: Prior to cycles 1, 4, 7, and 10 and then every 6 cycles thereafter, approximately 5 years
Population: Five patients were not analyzed due to clinical progression (n=1), plexiform neurofibroma surgery (n=1), progression in a pre-existing brain tumor (n=1), and refusal of further therapy (n=2).
Measure: Count of Participants; unit: Participants
Groups:
- Pirfenidone: Pirfenidone orally as capsules three times a day approximately every 8 hours for cycles of 28 days with no rest period between cycles (28 day treatment cycles); 500 mg/m^2 every 8 hours (1500 mg/m^2/day).
Arm/Group | Pirfenidone
Number analyzed (Participants) | 31
Participants
  Progressive disease | 31
  Complete response | 0
  Partial response | 0
  Stable disease | 0
  MInor response | 0

9. Secondary Outcome: Number of Participants Who Contributed to the Tissue Bank
Description: Tumor specimens from patients who undergo tumor surgery or biopsies for clinical reasons.
Time Frame: 5 years
Population: Participants declined to contribute specimens for the tissue bank.
Arm/Group | Pirfenidine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Pirfenidone
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 3/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=36)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=36)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (2)
Albumin, serum low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (7)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 7 (8)
Anorexia (Gastrointestinal disorders) | 9 (22)
Atrophy, skin (Skin and subcutaneous tissue disorders) | 1 (1)
Bicarbonate, serum low (Investigations) | 4 (7)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 4 (5)
Calcium, hypocalcemia (Metabolism and nutrition disorders) | 9 (13)
Cardiac arrhythmia-Other, specify- sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac general, Other-(specify-fluid retention) (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Constitutional symptoms (Other, specify-cold symptoms) (General disorders) | 3 (4) — cough insomnia
Dehydration (Gastrointestinal disorders) | 3 (3)
Dental: teeth (Gastrointestinal disorders) | 1 (1)
Dermatology/Skin-Other (Specify-multiple bug bites) (Skin and subcutaneous tissue disorders) | 4 (6) — nodule in L scapula rash caused by fungal infection cut foot 3 stitches insect bites
Diarrhea (Gastrointestinal disorders) | 21 (63)
Dizziness (Nervous system disorders) | 4 (5)
Dry eye syndrome (Eye disorders) | 1 (1)
Edema: head and neck (General disorders) | 1 (1)
Edema: limb (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 11 (21)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 10e9/L) (General disorders) | 10 (20)
Flu-like syndrome (General disorders) | 6 (7)
Gastrointestinal-Other (Specify- 1 episode of incontinence of bowel) (Gastrointestinal disorders) | 2 (2) — gastrointestinal-other, specify, stool, green
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4)
Glucose, serum low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 5 (10)
Hemorrhage, GU: Ovary (Reproductive system and breast disorders) | 1 (1)
Hemorrhage, GU: urinary NOA (Renal and urinary disorders) | 1 (2)
Hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypertension (Vascular disorders) | 3 (3)
Incontinence, urinary (Renal and urinary disorders) | 2 (2)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils (ANC < 1.0 x 10 (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils (ANC < 1.0 x 10e9/L: External ear (otitis externa)
Infection-Other (specify-infection) (Infections and infestations) | 6 (7) — infection oral cavity, thrush sinus infection sinus infection + cough bronchitis, congestion infection-ear
Leukocytes (total WBC) (Investigations) | 8 (22)
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (3)
Lymphatics-Other (Specify-bilateral lymphadenopathy) (Blood and lymphatic system disorders) | 4 (4) — lymphatics-other (specify-cervical lymphadenopathy) snoring and gasping shotty lymphadenopathy cervical chain
Lymphopenia (Blood and lymphatic system disorders) | 6 (8)
Magnesium, serum high (hype (Metabolism and nutrition disorders) | 8 (9)
Magnesium, serum low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3)
Mood alteration: agitation (Nervous system disorders) | 2 (2)
Mood alteration: depression (Nervous system disorders) | 2 (3)
Mucositis/stomatitis (clinical exam): oral cavity (Gastrointestinal disorders) | 2 (3)
Muscle weaknesses, generalized or specific area (not due to neuropathy): extreme-lower (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 29 (157)
Neurology-Other (specify-tic, constant clearing of throat) (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 7 (24)
Obstruction/stenosis of airway: bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstruction/stenosis of airway: larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ocular/Visual-Other (Specify-blurred vision intermittent) (Eye disorders) | 2 (2)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 3 (6)
PTT (partial thromboplastin time) (Investigations) | 1 (1)
Pain: abdomen NOS (Reproductive system and breast disorders) | 5 (8)
Pain: back (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain: bladder (Renal and urinary disorders) | 1 (3)
Pain: bone (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain: buttock (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: chest wall (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain: chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain: dental/teeth/peridontal (Gastrointestinal disorders) | 2 (3)
Pain: esophagus (Gastrointestinal disorders) | 1 (1)
Pain: extremity-limb (Musculoskeletal and connective tissue disorders) | 7 (13)
Pain: head/headache (Nervous system disorders) | 21 (52)
Pain: joint (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain: middle ear (Ear and labyrinth disorders) | 1 (1)
Pain: muscle (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain: neck (Musculoskeletal and connective tissue disorders) | 5 (15)
Pain: pain NOS (Nervous system disorders) | 4 (4)
Pain: pelvis (Reproductive system and breast disorders) | 1 (1)
Pain: penis (Reproductive system and breast disorders) | 1 (1)
Pain: skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: stomach (Gastrointestinal disorders) | 2 (2)
Pain: throat/pharynx/larynx (Gastrointestinal disorders) | 4 (5)
Personality/behavioral (Psychiatric disorders) | 5 (7)
Phosphate, serum low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3)
Platelets (Investigations) | 3 (5)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum low (hypokalemia) (Metabolism and nutrition disorders) | 4 (6)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 5 (7)
Pulmonary/upper respiratory-Other (Specify-bloody nose) (Respiratory, thoracic and mediastinal disorders) | 3 (5) — nasal congestion cold symptoms wheezing secondary to tracheitis
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (3)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Supraventricular and nodal arrhythmia: sinus tachycardia (Cardiac disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular-Other (Specify-vascular other specify, coolness LL) (Vascular disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (119)
Flushing (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Pain-Other (Specify-left ear pain) (Ear and labyrinth disorders) | 4 (6) — mild mouth aching orthodontic discomfort pain (head site of surgery) pain rt side
AST, SGOT (serum oxaloacetic transaminase) (Investigations) | 2 (3)
Alkaline phosphatase (Investigations) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils : bronchus (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : catheter-related (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : conjunctiva (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : foreign body (e.g. graft, implant, prosthesi (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : middle ear (otitis media) (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : penis (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : pharynx (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : sinus (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils : skin (cellulitis) (Infections and infestations) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils : upper aerodigestive NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils : upper airway NOS (Infections and infestations) | 5 (7)
Infection with unknown ANC : external ear (otitis externa) (Infections and infestations) | 2 (3)
Infection with unknown ANC : lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC : sinus (Infections and infestations) | 2 (2)
Infection with unknown ANC : trachea (Infections and infestations) | 1 (1)
Infection with unknown ANC : upper airway NOS (Infections and infestations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2008-04-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT00076102/Prot_SAP_ICF_000.pdf